CLINICAL TRIAL: NCT03021889
Title: Nutritional Therapy Improves Dyslipidemia in HIV Infected Teenagers With Antiretroviral Treatment: a Randomized Controlled Trial
Brief Title: Nutritional Therapy Improves Dyslipidemia in HIV Infected Teenagers With Antiretroviral Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 150018
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Adolescent Behavior; Hiv; Dyslipidemias
Keywords: HIV / AIDS; Dyslipidemia; Adolescents; Nutritional Therapy
MeSH Terms: conditions — Adolescent Behavior; Acquired Immunodeficiency Syndrome; Dyslipidemias | interventions — Nutrition Therapy; Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional therapy group (Experimental): The group nutritional therapy intervention was subjected to a protocol that included: nutritional counseling and weekly phone calls for 12 weeks.
  Interventions: Behavioral: Nutritional therapy
- Control group (Other): The control group received conventional care consisting of usual medical care. The control group was followed according to the ambulatory care routine, which consists of medical follow-up by the assistant team.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Nutritional therapy — The nutritional therapy intervention group received monthly nutritional guidelines for 12 weeks focusing on the diet for dyslipidemia, based on the recommendation of the type I diet of the Clinical Protocol and Therapeutic Guidelines for Management of HIV Infection in children and adolescents. In addition, participants in the intervention group received weekly phone calls for nutritional counseling.
  Arms: Nutritional therapy group
Behavioral: Control group — The control group was followed according to the ambulatory care routine, which consists of medical follow-up by the assistant team.
  Arms: Control group

SUMMARY:
Introduction: Prolonged use of antiretroviral therapy is associated with metabolic and bodily changes such as lipodystrophy, diabetes mellitus, insulin resistance and dyslipidemia latter being associated with a higher chance of cardiovascular events and death.

Objective: To evaluate the effect of nutritional therapy in dyslipidemic adolescents living with HIV / AIDS in antiretroviral therapy.

Method: This is a randomized clinical trial with young people 13-19 years in outpatient treatment in a general hospital to present dyslipidemia. The intervention group received nutritional counseling for 12 weeks and weekly flights to nutritional counseling. The control group received standard care consisting of medical care. Demographic, clinical, nutritional variables, food surveys and lipid profiles were collected at baseline and at the end of the study for both groups.

DETAILED DESCRIPTION:
This is a open randomized clinical trial. The participants were adolescents (13 to 19 years old) diagnosed with HIV / AIDS from the Pediatric Infectious Disease Outpatient Clinic - zone 4, from a tertiary care university hospital in the South Region in Brazil, along with their caregivers. Present Dyslipidemia, characterized by Total Cholesterol> 200mg / dL associated with:Triglycerides ≥ 150mg HDL cholesterol (male <40 mg / dL and female <50 mg / dL) LDL cholesterol ≥ 160 mg / dL. The clinical profile, immunological, virological, the biochemical parameters will be accessed by the patient's chart and the dietary parameters will be evaluated by means of 24-hour reminder instrument. The sample was calculated, using a software, from an alpha error of 5%, reliability power of 80%, to obtain detection difference and standard deviation for each of the group of 40, totaling 36 patients.

The randomization will be performed through simple randomization in blocks of 2 patients generated by computer program, available at www.randomization.com.

The intervention group received nutritional counseling for 12 weeks and weekly flights to nutritional counseling. The control group received standard care consisting of medical care. Demographic, clinical, nutritional variables, food surveys and lipid profiles were collected at baseline and at the end of the study for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HIV infection with a positive result obtained by performing a screening test for anti-HIV-1 and anti-HIV-2 and at least one confirmatory test;
* Being on antiretroviral therapy for at least three months prior to the start of the study;
* Present current biochemical exams: Dyslipidemia, characterized by Total Cholesterol> 170mg / dL associated with: Triglycerides greater than or equal to LDL cholesterol ≥ 130 mg / dL;
* Availability to participate in the nutritional intervention with a low fat diet.

Exclusion Criteria:

* Pregnant women;
* Patients with active opportunistic infections;
* Cognitive deficits;
* Diabetes mellitus;
* Patients taking lipid-lowering drugs;
* Patients who are unaware of their HIV diagnosis.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Blood plasma level of total cholesterol | 12 months
  Total blood cholesterol level will be assessed by blood test

SECONDARY OUTCOMES:
Food intake | 12 months
  Food intake will be assessed a 24-hour reminder
Nutritional status | 12 months
  Will be assessed by body mass index
Blood plasma level of triglycerides | 12 months
  Triglycerides level will be assessed by blood test
Blood plasma level of HDL cholesterol | 12 months
  HDL cholesterol level will be assessed by blood test

CONTACTS AND LOCATIONS:
Overall Officials: Michelli S de Assis, PhD, Principal Investigator — Nurse Research

IPD SHARING:
Plan to Share IPD: Undecided